CLINICAL TRIAL: NCT01529580
Title: School-Age Children With Autism With Limited Expressive Language Skills: An Intervention Study
Brief Title: School-Age Children With Autism With Limited Expressive Language Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca Landa, Director of the Center for Autism and Related Disorders (CARD) and Professor, Johns Hopkins University School of Medicine, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00049467; 3R01MH085048-03S1 (NIH)
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; language; intervention; school-age
MeSH Terms: conditions — Autism Spectrum Disorder; Language | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 Week Basline Prior to Intervention (Experimental): If eligible, you will be randomly assigned- as if by flipping a coin- to one of three baseline durations, during which your child will engage in daily interactions with their interventionist to determine if skills targeted by this intervention are improving naturally as your child matures, without active treatment from the study's interventionist. In this case, the duration is 1 week before your child begins active treatment with their interventionist.
  Interventions: Behavioral: Non-Verbal School Aged Children with Autism (NVSACA) Intervention
- 2 Week Basline Prior to Intervention (Experimental): If eligible, you will be randomly assigned- as if by flipping a coin- to one of three baseline durations, during which your child will engage in daily interactions with their interventionist to determine if skills targeted by this intervention are improving naturally as your child matures, without active treatment from the study's interventionist. In this case, the duration is 2 weeks before your child begins active treatment with their interventionist.
  Interventions: Behavioral: Non-Verbal School Aged Children with Autism (NVSACA) Intervention
- 3 Week Basline Prior to Intervention (Experimental): If eligible, you will be randomly assigned- as if by flipping a coin- to one of three baseline durations, during which your child will engage in daily interactions with their interventionist to determine if skills targeted by this intervention are improving naturally as your child matures, without active treatment from the study's interventionist. In this case, the duration is 3 weeks before your child begins active treatment with their interventionist.
  Interventions: Behavioral: Non-Verbal School Aged Children with Autism (NVSACA) Intervention

INTERVENTIONS:
Behavioral: Non-Verbal School Aged Children with Autism (NVSACA) Intervention — The intervention has 3 components:
  1. One-on-one play based intervention: administered by the interventionist at the school for 1 hour, three times a week, each week for the 5 month duration of the intervention.
  2. Parent training: at the beginning of the 5th month of intervention, parents will receive training once a week for an hour during the remaining four weeks of intervention.
  3. Teacher training: in month 2 of the intervention, the teacher will receive 2 1.5 hour training sessions along with a weekly in-class coaching given as needed following completion of the second session of training.

SUMMARY:
This project will address a major challenge to the field of autism research: improving expressive communication in children with autism who have reached school age but have not acquired functional spoken language (non-verbal school aged children with autism; NVSACA).

Fifteen children who completed the RO1 ICAN intervention (NCT01018407) at the Kennedy Krieger site and follow-up testing but continue to have minimal functional spoken language will be participants in this study. After eligibility is established, participants will be randomly assigned to a baseline duration of one week, two weeks or three weeks before the start of active treatment. Once the baseline duration is completed, participants begin active treatment one hour of intervention three days per week in the participants' school setting. In month 2, weekly teacher trainings begin. In month 5, weekly parent trainings begin to improve the child's generalization of skills and teach parents the strategies implemented in their child's treatment. Post-baseline and post-treatment assessments will be completed in the lab at a time that is convenient for the participants' families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism by a licensed psychologist or board certified developmental pediatrician, or child and adolescent psychiatrist, confirmed by the Autism Diagnostic Observation Schedule (ADOS; Lord, Rutter, DiLavore, & Risi, 1999)
* Chronological age between 4.0 years and 7 years, 11 months
* Reynell developmental score ≤ 24 months, ADOS A1 score of 2, 3 or 8
* Nonverbal IQ of ≥ 40 (Leiter International Performance Scale-Revised (Leiter-R), Roid & Miller, 2007)
* Children have participated in and completed follow-up testing for the ICAN study.

Exclusion Criteria:

* Major medical conditions other than autism (e.g., genetic disorders [e.g., Fragile X, Down syndrome, tuberous sclerosis], blindness or deafness, and motor disabilities such as cerebral palsy;
* Uncontrolled seizures;
* Self-injurious behavior or moderate to severe aggression.
* Children in foster care.
* Children who are exposed to < 50% English throughout their typical day.
* Children currently participating in another intervention/treatment study.

Ages: 48 Months to 95 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Spontaneous Language | Weekly throughout the 5 month intervention (baseline and 5 months)
  The number of unprompted spontaneous language during a 15min play sample.

SECONDARY OUTCOMES:
Change in Baseline Autism Diagnostic Observation Schedule | 5 months into treatment (at completion of intervention)
Change in Baseline Reynell | 5 months into treatment (at completion of intervention)
Changes in Baseline Early Social Communication Scales (ESCS) | 5 months into treatment (at completion of intervention) and 6 months following the completion of the intervention
Changes in Baseline Structured Play Assessment | 5 months into treatment (at completion of intervention) and 6 months following the completion of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, CCC-SLP, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States